CLINICAL TRIAL: NCT00936845
Title: Females With Severe or Moderate Hemophilia A or B: A Multi-Center Study
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: CSL Behring (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: Females with Hemophilia
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Females with Hemophilia: Females with severe or moderate Hemophilia A or B.

SUMMARY:
To collect and analyze data on females with hemophilia so as to better define the difference between the study population and the male population with hemophilia.

DETAILED DESCRIPTION:
This study is designed as an epidemiological study with retrospective clinical and genetic data collection and prospective quality of life (QOL) data collections and genotyping of subjects without current molecular diagnosis. Data on the genetic/chromosomal etiology of the condition will be collected through chart review. For those subjects who have not had molecular or cytogenetic analysis, molecular and cytogenetic testing will be offered after genetic counseling. Those subjects who agree to have genetic testing will have 5-10 ml of blood drawn and sent to the cytogenetic laboratory at Weill Cornell Medical College for testing to determine the chromosomal complement, and 5 ml of blood sent to Dr. Arupa Ganguly at the University of Pennsylvania for the identification of a factor VIII or factor IX mutation, and X-chromosome inactivation studies.

ELIGIBILITY:
Inclusion Criteria:

* Females with severe (FVIII<0.01u/dl) or moderate (FVIII-0.01<0.06 u/dl) hemophilia A
* Females with severe (FIX<0.01u/dl) or moderate (FIX-0.01<0.06u/dl) hemophilia B
* Willingness to participate in the study.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria with respect to gender or hemophilia severity.

Min Age: 1 Month | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females with severe or moderate (less than 5%) hemophilia A or B.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2005-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of females with severe or moderate hemophilia A or B in the United States. | Study Duration

SECONDARY OUTCOMES:
Collect existing data on the genetic and/or chromosomal causes for severe and moderate hemophilia A and B in females in the United States. | Study Duration
To determine the natural history of hemophilia in females by collecting and analyzing data on the symptoms, treatment patterns, and complications of hemophilia in this cohort. | Study Duration
Collect and analyze data on the health-related quality of life and psychosocial adaptation to disease of females in the United States. | Study Duration

CONTACTS AND LOCATIONS:
Overall Officials: William B Mitchell, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (19):
- United States (18):
  - City of Hope National Medical Center, Duarte, California
  - Mountain States Regional Hemophilia and Thrombosis Center, Aurora, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hemophilia Program Office, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky Hemophilia Treatment Center, Lexington, Kentucky
  - Boston Hemophilia Center- Children's Hospital, Boston, Massachusetts
  - Henry Ford Hospital Adult Hemophilia and Thrombosis Treatment Center, Detroit, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Hemophilia Center of Western New York - Pediatric, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - Mary M. Gooley Hemophilia Center, Inc., Rochester, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oklahoma Center for Bleeding Disorders, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
- Puerto Rico Hemophilia Treatment Center, San Juan, Puerto Rico